CLINICAL TRIAL: NCT05626257
Title: Regulatory Post-Marketing Surveillance (rPMS) of Xolair® (Xolair® 150mg Powder for Solution for Injection, Xolair® 150mg/1ml Liquid in Pre-filled Syringe, Xolair® 75mg/0.5ml Liquid in Pre-filled Syringe) for Chronic Rhinosinusitis With Nasal Polyps (CRSwNP)
Brief Title: Regulatory Post-Marketing Surveillance of Xolair® for Chronic Rhinosinusitis With Nasal Polyps
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CIGE025EKR04
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps
Keywords: Chronic Rhinosinusitis with Nasal Polyps; CRSwNP; Korea; NIS; Xolair
MeSH Terms: interventions — Omalizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Xolair: patients who prescribed with Xolair according to the current label information in Korea.
  Interventions: Other: Xolair

INTERVENTIONS:
Other: Xolair — There is no treatment allocation. Patients administered Xolair by prescription that have started before inclusion of the patient into the study will be enrolled.

SUMMARY:
This study aims to evaluate the safety and effectiveness of Xolair® in patients with chronic rhinosinusitis with nasal polyps in routine clinical practice.

DETAILED DESCRIPTION:
This is a 24-week, prospective, open-label, multi-center, single-arm, observational, post-marketing surveillance study under routine clinical practice and does not impose a therapy, visit, or assessment. The study design was approved by the Korean health authority. The purpose of this study is not to answer scientific hypotheses, but to describe the incidences of all potential adverse events (AEs), serious adverse events (SAEs), and unexpected AEs not listed in the local label information occurring in Korean patients under routine clinical practice following the approved local label information.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged ≥18 years
2. Patients with CRSwNP who are not adequately controlled with conventional therapy (INCS)
3. Patients prescribed with Xolair® as per the locally approved label information.
4. Patients who provide written informed consent to participate in the study

Exclusion Criteria:

1. Patients who do not provide consent to participate in the study
2. Patients participating in other clinical trial
3. Contraindications listed in the locally approved label information of Xolair®

   * Hypersensitivity to the active ingredient or any other ingredient of Xolair®
   * Patients with myocardial infarction or history of myocardial infarction (pre-filled syringes only)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: this study will involve patients who received at least one dose of Xolair® for the treatment of Chronic Rhinosinusitis with Nasal Polyps (CRSwNP) according to the current label information in Korea.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Incidences of adverse events/adverse drug reactions (AEs/ADRs) | Up to 24 weeks
  Incidences of adverse events/adverse drug reactions (AEs/ADRs), serious AEs/ADRs (SAEs/SADRs), unexpected AEs/ADRs (UAEs/UADRs), serious unexpected AEs/ADRs (SUAEs/SUADRs) will be collected

SECONDARY OUTCOMES:
Change from baseline in SNOT-22 | Baseline, Week 12 and Week 24
  Sino-Nasal Outcome Test-22 (SNOT-22) is a validated questionnaire that is used to assess the impact of chronic rhinosinusitis on health-related quality of life (HRQoL). It is a 22 item questionnaire with each item assigned a score ranging from 0 (no problem) to 5 (problem as bad as it can be). The total score may range from 0 (no disease) to 110 (worst disease), lower scores representing better health related quality of life.
Incidences of AEs by subject characteristics | Up to 24 weeks
  The incidences of AEs by subject characteristics (demographic and other baseline information, Xolair® administration status, concomitant medication and therapy, etc.). The significance of the difference in the incidence of adverse events between categories within each characteristic will be tested using the Chi-square test or Fisher's exact test.
Subject characteristics that affect the occurrence of adverse events | Up to 24 weeks
  Logistic regression analysis will be performed to analyze subject characteristics that affect the occurrence of adverse events.
change from baseline in SNOT-22 according to subject characteristics | Week 12 and Week 24
  Change from baseline in SNOT-22 according to subject characteristics (demographic and other baseline information, Xolair® administration status, concomitant medication and therapy, etc.). The statistical significance of the difference in the change between the groups will be tested by two-sample t-test, Wilcoxon rank sum test, ANOVA, or Kruskal-Wallis test.
Subject characteristics that affect the change from baseline in SNOT-22 | Week 12 and Week 24
  Multivariate linear regression analysis will be performed to evaluate the subject characteristics (demographic and other baseline information, Xolair® administration status, concomitant medication and therapy, etc.) that affect the change from baseline in SNOT-22

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- South Korea (10):
  - Novartis Investigative Site, Anyang-si, Gyeonggi-do
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Uijeongbu-si, Gyeonggi-do
  - Novartis Investigative Site, Incheon, Korea
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Yangcheon gu
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Gyeonggi-do
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Suwon

IPD SHARING:
Plan to Share IPD: No